CLINICAL TRIAL: NCT07332299
Title: Remote Stimulation and Training to Advance Recovery From TBI in Seniors
Acronym: ReSTART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Center for Veterans Research and Education (Other)
Responsible Party: Principal Investigator, Casey Gilmore, PhD, Principal Investigator, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1893132; SCI-TBI-2025-00025 (Other Grant/Funding Number: State of Minnesota Office of Higher Education)
Record Dates: First submitted 2025-09-17; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Traumatic Brain Injury; Aging Related Cognitive Decline
Keywords: Aging; Cognitive Training; Transcranial Direct Current Stimulation; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active tDCS with cognitive training (Experimental): Participants will receive 10 sessions of cognitive training concurrent with transcranial direct current stimulation (45 minutes of cognitive training with tDCS applied for first 20 minutes of session; tDCS: 2mA, 30s ramp up/down, anode at F3, cathode at F4).
  Interventions: Combination Product: Active tDCS and Cognitive Training Intervention
- Sham tDCS with cognitive training (Sham Comparator): Participants will receive 10 sessions of cognitive training concurrent with sham transcranial direct current stimulation (45 minutes of cognitive training with sham tDCS: 2mA current will be ramped down immediately after the initial 30s ramp up period and then at 20 minutes ramped up and down as done at the beginning, anode at F3, cathode at F4).
  Interventions: Combination Product: Sham tDCS and Cognitive Training Intervention

INTERVENTIONS:
Combination Product: Active tDCS and Cognitive Training Intervention — Forty-five minutes of cognitive training concurrent with 2 mAmps of anodal stimulation applied to the left frontal cortex for the first 20 minutes of the session.
  Other Names: tDCS
  Arms: Active tDCS with cognitive training
Combination Product: Sham tDCS and Cognitive Training Intervention — Forty-five minutes of cognitive training concurrent with sham tDCS (30 secs ramp up/ramp down of current at beginning and end of session).
  Other Names: sham tDCS
  Arms: Sham tDCS with cognitive training

SUMMARY:
The goal of this clinical trial is to learn if combining brain stimulation with cognitive training can improve thinking skills in older adults who have had a traumatic brain injury (TBI).

The main questions are:

* Does transcranial direct current stimulation (tDCS) make cognitive training more effective for improving attention, memory, and decision-making?
* Is this type of home-based program feasible and acceptable for older adults with TBI?

Researchers will compare two groups: one group will receive active tDCS during cognitive training, and the other group will receive sham (placebo) tDCS during cognitive training.

Participants will:

* Complete computer-based cognitive training exercises (BrainHQ) to practice attention, memory, and decision-making.
* Receive either active or sham tDCS during training sessions.
* Complete assessments before and after the program to measure changes in thinking and daily functioning.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a major public health issue among older adults. Each year, thousands of seniors sustain TBIs, most often from falls. Even when the injury is classified as "mild," it can lead to long-term problems with memory, attention, decision-making, and self-control. These difficulties can make it harder to live independently, maintain social relationships, and manage everyday responsibilities. Older adults with a history of TBI are also at greater risk of experiencing faster cognitive decline as they age. Unfortunately, there are few effective treatments available to improve thinking skills in this group.

This study is designed to test a new approach that combines **computer-based cognitive training** with **transcranial direct current stimulation (tDCS)**, a safe, non-invasive form of brain stimulation. The goal is to determine whether this combined treatment can improve attention, memory, and decision-making in older adults with TBI, and whether the program is practical for participants to complete at home with remote supervision.

About the Interventions

* Cognitive training (BrainHQ): Participants will complete computerized exercises that provide structured practice in skills such as attention, working memory, and decision-making. These exercises adapt to each individual's performance, gradually increasing in difficulty as skills improve.
* tDCS: During some of the training sessions, participants will wear a device with electrodes placed on the scalp. The device delivers a very low level of electrical current (2 milliamps) that helps "tune" brain networks to make them more responsive to training. tDCS is non-invasive, painless for most people, and has been tested safely in thousands of participants in research studies worldwide.

Study Design

This is a randomized controlled trial. All participants will complete the same set of cognitive training exercises, but they will be randomly assigned to one of two groups:

* Active group: Receives active tDCS during training.
* Sham group: Receives sham (placebo) tDCS during training. Sham stimulation mimics the feeling of tDCS at the start of the session but does not deliver active current.

This design allows researchers to determine whether adding tDCS produces greater improvements than cognitive training alone.

Study Procedures

Participants will:

1. Complete baseline assessments of cognitive function, daily living skills, and quality of life.
2. Take part in multiple sessions of computer-based cognitive training at home, while supervised remotely through secure telehealth connections.
3. Receive either active or sham tDCS during the training sessions.
4. Complete follow-up assessments after the intervention to measure changes in thinking, decision-making, and daily functioning.

Key Questions

The study is designed to answer three main questions:

1. Does tDCS enhance the effects of cognitive training? Specifically, do participants who receive active tDCS show greater gains in attention, memory, and decision-making compared to those who receive sham stimulation?
2. Is the program feasible and acceptable? Can older adults with TBI successfully complete the home-based training and stimulation sessions, and do they find the program easy to use and worthwhile?
3. Do improvements transfer to everyday life? Beyond test scores, does the program help participants function better in their daily lives, maintain independence, and improve quality of life?

Importance of the Study

Older adults with TBI are at particularly high risk for poor outcomes, but they are often underrepresented in research. This study is innovative in several ways:

* It focuses specifically on older adults with TBI, a group that has historically been overlooked in clinical trials.
* It uses a home-based and remotely supervised model, which increases accessibility for people living in rural areas, those with mobility limitations, or those who cannot easily attend clinic visits.
* It builds on strong preliminary evidence from prior studies in Veterans and other populations showing that combining brain stimulation with cognitive training can reduce impulsivity and improve cognitive control.
* It addresses a critical gap in treatment by testing a scalable rehabilitation approach that could be delivered widely if proven effective.

Potential Impact

If successful, this research could provide the foundation for a new, effective treatment option for older adults with TBI. The intervention is low-risk, non-invasive, and can be delivered in the home setting with minimal equipment. It could help participants improve cognitive functioning, maintain independence longer, and enhance quality of life. At a broader level, the study could reduce the burden of TBI-related cognitive decline on families, caregivers, and healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

1. Veterans age 65 and older.
2. History of mild TBI (as defined by the DOD/VA criteria used in conjunction with the OSU TBI-ID) sustained at least 3 months prior to enrollment.
3. Self-reported or medically documented attention and/or concentration difficulties.
4. Stable dose of all prescription and non-prescription medications that may impact cognition or brain chemistry (except for PRN medication) for at least 3 weeks prior to the baseline session (Visit 1), in the medical opinion of the principal investigator.
5. Capable and willing to provide voluntary informed consent, in the medical opinion of the principal investigator.

Exclusion Criteria:

1. Presence of a medical, psychiatric, physical or non-physical disease, disorder, condition, injury, disability or pre-existent history such that study participation, in the opinion of the principal investigator: (a) may pose a significant risk to the participant, (b) raises the possibility that the participant is unlikely to successfully complete all the requirements of the study according to the study protocol, or (c) might adversely impact the integrity of the data or the validity of the study results. Specific conditions include (but are not limited to) a history of brain tumor near the stimulation site, brain surgery, stroke with current sequalae, epilepsy, multiple sclerosis, Huntington's Disease, ALS, ataxia, aphasia, Alzheimer's Disease, and dementia.
2. Moderate to severe cognitive impairment with MoCA score (assessed upon enrollment) less than 15.
3. Prior treatment with ECT or neuromodulation in the last 12 months.
4. Current severe alcohol or substance use disorder with evidence of withdrawal or tolerance within the past 6 months, based on psychiatric history and/or a review of available medical records.
5. Psychosis or mania within 30 days of enrollment, as determined by the principal investigator, based on psychiatric history and/or a review of available medical records.
6. Contraindications for tDCS (e.g., metallic cranial plates/screws or implanted device, eczema or skin lesions on scalp near electrode site, etc.).
7. No or limited internet connection in their home.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Total Scale Score | Baseline, 1-week post, & 6-weeks post intervention
  The RBANS is a commonly-used, psychometrically-sound measure of cognitive function across the lifespan. The primary outcome measure is the Total Scale score, which is a standard score (mean 100, SD 15) across five cognitive domains (Immediate/Delayed Memory, Visuospatial, Attention, Language).
Electroencephalogram (EEG) - Resting State Theta Band Functional Connectivity | Baseline, 1-week post, & 6-weeks post intervention
  Resting State EEG will be collected to assess neural dynamics or functional connectivity and spectral power of delta,theta, alpha, beta, and gamma frequency bands. The primary outcome measure will be change in prefrontal-parietal functional connectivity in the theta frequency band.

SECONDARY OUTCOMES:
Neurobehavioral Symptom Inventory (NSI) Total Score | Baseline, 1-week post, & 6-weeks post intervention
  A 22-item measure that assesses post-concussive symptoms for those with a TBI.
Insomnia Severity Index (ISI) Total Score | Baseline, 1-week post, & 6-weeks post intervention
  A 7-item measure of the severity of nighttime and daytime components of insomnia.
Patient Health Questionnaire-8 (PHQ-8) Total Score | Baseline, 1-week post, & 6-weeks post intervention
  An 8-item measure of depressive symptoms.
Groton Maze Learning Task (GMLT) Completion Time | Baseline, 1-week post, & 6-weeks post intervention
  A computer cognitive test of spatial working memory and error monitoring.
NIH Toolbox Quality of Life Assessment (NeuroQoL) | Baseline, 1-week post, & 6-weeks post intervention
  Questionnaire to assess quality of life with regard to cognitive, social, emotional, and behavioral abilities.

CONTACTS AND LOCATIONS:
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No